CLINICAL TRIAL: NCT03328637
Title: Smartphone Addiction and Its Effect on Mental Health: An Evidence Based Intervention for Amelioration
Acronym: CyberLife Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University, Islamabad (Other)
Responsible Party: Principal Investigator, Muhammad Tahir Khalily, Professor, International Islamic University, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11/09/17-P01-DPEC
Record Dates: First submitted 2017-10-04; First posted 2017-11-01 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Smartphone Addiction
Keywords: Smartphone Addiction; CBT; Evidence based intervention
MeSH Terms: conditions — Internet Addiction Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The study is a Randomized Controlled Trial (RCT) with single blind rating. The randomization of participants is across two groups (1) one provided with intervention of CBT and (2) the other group will be on Treatment As Usual (TAU)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group will be provided Cognitive Behavioral Therapy (CBT). CBT is a common psychological intervention based on the notion that thoughts trigger the emotions. In CBT patients are trained to monitor their thoughts and identify those that trigger addictive feelings and actions while they learn new coping skills and ways to prevent a relapse (Beck, Wright, Newman & Liese, 2001). The treatment period of CBT is three months consisting of a weekly session and total 12 sessions. Initial stage of therapy is behavioral, centering on specific behaviors and situations. Latter on there is more of a focus on the cognitive assumptions and distortions that have developed and the effects of these on behavior.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Control (No Intervention): Control group will not receive CBT however, primary care service providers and mental health professionals will provide any required routine care according to their clinical judgment and available resources.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT) consisting of weekly 12 sessions will focus on moderated and controlled use of smartphone instead of abstinence model.
  Arms: Intervention

SUMMARY:
The use of Smartphone has been adopted faster than any other device in the history of digital electronics. Hence it is estimated that in 2016, 2.1 billion were found registered Smartphone users in the world and Pakistan was ranked 10th in the list of top 10 countries with largest number of mobile phone subscribers. Despite of its useful and timely utilization, the excessive use of Smartphone coerce the Individual to be dependent on the use of Smartphone psychologically and even physically. Furthermore, among the users, adolescents and young adults used Smartphone (90%) more than any other age groups. Moreover, this prevalence is expected to rise in the future due to the easy availability and swift changes and addition of new applications to Smartphone technology. Subsequently, the excessive and irrational use of Smartphone leads to Smartphone addiction which impact on individual mental health, physical health, and disrupt social, economic and educational functions. So, this study aims to assess the effectiveness of Cognitive Behavioral Therapy (CBT) as an evidence based remedy in the treatment of Smartphone addiction. The study will comprise of two groups; one will receive CBT (intervention group) and the other one will be on Treatment As Usual (TAU). The aim of the study is to assess the effectiveness of CBT primarily by measuring the addictive smartphone usage assessed by Smart Phone Addiction Scale (SAS) and also on secondary outcomes including time management, academic performance and social functioning of adolescents. These assessments will be conducted before intervention (on the baseline assessment sessions), during the Intervention and after the intervention (on follow up assessment sessions). A total of 120 students were calculated on the basis of 80% statistical power required to detect the effect as indicated by previous study and will be selected from different educational institutions. SPSS 23.0 will be used for data analysis. The primary analysis will be mixed ANOVA to compare the between group and within group means differences on measures used in the study. Multiple Hierarchical Regression analysis will also be used for the prediction of outcome variables from the demographics. The total duration of the study is one year.

This study primarily aims to assess the effectiveness of Cognitive Behavioral Therapy (CBT) as an evidence based remedy in the treatment for Smartphone addiction. The basic purpose is to minimize the severity of Smartphone addiction up to manageable level. Furthermore, there are certain psychiatric symptoms that are found to be associated with the addictive usage of Smartphone like stress, depression, anxiety, hyperactivity, attention deficits and conduct problems. The study design will also allow to assess the effectiveness of CBT on such outcomes: (a) The depression, anxiety and stress level of the participants (b) The time management of the participants (c) The emotional symptoms, conduct problems, hyperactivity and attention deficit problems, peer relationship problems and pro-social behavior aspects of the participants (d) The satisfaction level of the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Score more than 31 (for male) and 33 (for female) on Smart Phone Addiction Scale Short Version (SAS-SV).
2. Age range will be 12-19.
3. Absence of diagnosis according to ICD-10 or DSM 5 mental disorder.
4. Participants will have to be living within the catchment area.
5. Capable to be engaged, participate or respond to the research question.
6. Willing to give informed consent.

Exclusion Criteria:

1. Temporary resident unlikely to be available for the follow ups.
2. Participants diagnosed according to ICD 10 or DSM 5 criteria, due to general medical condition or substance misuse, dementia, delirium, alcohol or drug dependence, schizophrenia, bipolar disorder, learning disability.
3. Unable to engage, participate or respond to the research question.
4. Participants who attended psychiatric services

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Smartphone Addiction Scale (SAS; Assessing Change) | Assessments will be conducted at baseline (after the screening), 6th week (1/2 month) after the baseline, 12th week (3rd month) after the baseline and at 6th month. The purpose of the outcome measure is to asses the change from baseline to follow-up.
  Smartphone Addiction Scale (SAS) is used to asses the severity of smartphone dependency and addiction. It consists of 33 items (Kwon et al., 2013). Individuals have to respond on the Likert scale between 1-6, where 1 indicates strongly disagree and 6 indicates strongly agree. The amounts of answers were divided to three levels of addiction: low (1-66), medium (67-132) and high (133-198). Internal reliability of SAS was found to be α = .99. This scale will be used as a primary outcome and will be included in the baseline and follow ups assessment to assess the degree of change from baseline to 3rd month and 6th month follow-ups.

SECONDARY OUTCOMES:
Depression Anxiety Stress Scales (DASS-42) | Assessments will be conducted at baseline (after the screening), 6th week (1/2 month) after the baseline, 12th week (3rd month) after the baseline and at 6th month.
  It is 42 items scale developed by Levibond and Levibond (1995). It has three subscales and each of them contains 14 items. The depression scale, the anxiety scale and the stress scale. There are cut off scores established to categorize the individual scores in the mild, moderate, severe, and extremely severe categories. It has 4-point rating scale ranging from 1 (Did not apply to me at all) to 4 (Applies to me most of the time). This questionnaire will be used in the baseline and follow-ups assessment sessions.
Strengths and Difficulties Questionnaire | Assessments will be conducted at baseline (after the screening), 6th week (1/2 month) after the baseline, 12th week (3rd month) after the baseline and at 6th month.
  This scale has 25 items in all and uses a 3 point Likert scale supporting five factors: 'emotional symptoms', 'conduct problems', 'hyperactivity and attention deficit problems', 'peer relationship problems' and 'prosocial behavior' (Goodman, 1997). For the first four factors, the lower the score, the better, and for the last factor the higher the score, the better. This question will be also used in the baseline and follow-ups assessment sessions.
Satisfaction with Life Scale (SWLC) | Assessments will be conducted at baseline (after the screening), 6th week (1/2 month) after the baseline, 12th week (3rd month) after the baseline and at 6th month.
  Satisfaction with Life Scale (SWLC) is a 5-item scale designed to measure the global cognitive judgements of one's life satisfaction (Diener, Emmons, Larsen & Griffin, 1985). Participants indicate how much they agree or disagree with each of the five items using a 7-point scale that ranges from 7 strongly agree to 1 strongly disagree. The higher score indicates higher satisfaction. This scale will be used in our baseline and follow-ups assessment sessions.
Client Satisfaction Questionnaire (CSQ) | The questionnaire will be employed on the 6th week (1/2 month) after the baseline, 12th week (3rd month) after the baseline and at 6th month
  The Client Satisfaction Questionnaire is a brief and simple scale to measure the patient satisfaction with mental health services (Gani, Saeed, Minhas, Anjuman, Waleed & Fatima, 2011). The questionnaire has 8 items and the participants have to respond on 4 point Likert scale ranging from 1 to 4. The total score of participant ranges from 8 to 32 where minimum score 8 reflects dissatisfaction and a maximum score 32 reflects maximum satisfaction. This questionnaire will be used after all of the intervention (CBT) sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychology, International Islamic University Islamabad Pakistan, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: SAP

REFERENCES:
- [Background] Kwon M, Kim DJ, Cho H, Yang S. The smartphone addiction scale: development and validation of a short version for adolescents. PLoS One. 2013 Dec 31;8(12):e83558. doi: 10.1371/journal.pone.0083558. eCollection 2013. PMID 24391787
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the Beck Depression and Anxiety Inventories. Behav Res Ther. 1995 Mar;33(3):335-43. doi: 10.1016/0005-7967(94)00075-u. PMID 7726811
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Gani N, Saeed K, Minhas FA, Anjuman N, Waleed M, Fatima G. Assessment of patient satisfaction with mental health services in a tertiary care setting. J Ayub Med Coll Abbottabad. 2011 Jan-Mar;23(1):43-6. PMID 22830144
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Wright FD, Beck AT, Newman CF, Liese BS. Cognitive therapy of substance abuse: theoretical rationale. NIDA Res Monogr. 1993;137:123-46. PMID 8289917
- [Derived] Khalily MT, Bhatti MM, Ahmad I, Saleem T, Hallahan B, Ali SA, Khan AA, Hussain B. Indigenously adapted cognitive-behavioral therapy for excessive smartphone use (IACBT-ESU): A randomized controlled trial. Psychol Addict Behav. 2021 Feb;35(1):93-101. doi: 10.1037/adb0000677. Epub 2020 Jul 23. PMID 32700919
- See also: Number of smartphone users worldwide from 2014 to 2020 (in billions) — http://www.statista.com/statistics/330695/number-of-smartphone-users-worldwide/